CLINICAL TRIAL: NCT01733745
Title: SYSTANE® Family Efficacy in Meibomian Gland Functionality for Lipid Deficient Evaporative Dry Eye Subjects
Brief Title: SYSTANE® Family - Meibomian Deficiency
Acronym: M-12-077
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A00978
Record Dates: First submitted 2012-11-21; First posted 2012-11-27 (Estimated); Results first posted 2014-07-03 (Estimated); Last update posted 2018-06-29 (Actual); Status verified 2013-09

CONDITIONS: Dry Eye Syndrome
Keywords: dry eye; lipid deficiency; meibomian gland
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SYSTANE® Family (Experimental): SYSTANE® Lid Wipes administered to treated eye(s) once a day; SYSTANE® BALANCE lubricant eye drops administered to treated eye(s), 1 drop 4 times a day; SYSTANE® Vitamins, 2 softgels ingested daily. Duration of treatment was 3 months.
  Interventions: Other: SYSTANE® Lid Wipes; Other: SYSTANE® BALANCE; Dietary Supplement: SYSTANE® Vitamins
- Standard of Care (Active Comparator): Microfiber towels (as warm compresses, with or without saline eye drops) warmed to the maximum comfortable temperature and placed over closed eyes for 8 minutes, 1 time a day. Duration of treatment was 3 months.
  Interventions: Other: Microfiber towels (as warm compresses, with or without saline eye drops)

INTERVENTIONS:
Other: SYSTANE® Lid Wipes — Pre-moistened eyelid cleansing wipes for topical ocular external scrubbing of eyelids and eyelashes
  Arms: SYSTANE® Family
Other: SYSTANE® BALANCE — Lubricant Eye Drops
  Arms: SYSTANE® Family
Dietary Supplement: SYSTANE® Vitamins
  Other Names: SYSTANE® Vitamin Omega-3 Supplement
  Arms: SYSTANE® Family
Other: Microfiber towels (as warm compresses, with or without saline eye drops)
  Arms: Standard of Care

SUMMARY:
The purpose of this study was to assess the efficacy of the SYSTANE® family of products (SYSTANE® Lid Wipes, SYSTANE® BALANCE Lubricant Eye Drops, and SYSTANE® Vitamins) on meibomian gland functionality in subjects with lipid deficiency related to evaporative dry eye as compared to the standard of care warm compresses.

ELIGIBILITY:
Inclusion Criteria:

* Must have a clinical diagnosis of lipid deficient Evaporative Dry Eye;
* Meibomian Gland Functionality - Not more than 6 glands yielding liquid secretion;
* Must be willing to discontinue the use of all other Meibomian Gland; Dysfunction management prior to receiving the study test article at Visit 1, up until the end of the study period;
* Must have best corrected visual acuity of 20/40 Snellen or better in each eye;
* Must be able to follow instructions and be willing and able to attend required study visits;
* Must read, sign, and date an Ethics Committee reviewed and approved informed consent form;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* History or evidence of ocular or intraocular surgery or serious ocular trauma in either eye within the past 6 months;
* Current punctal occlusion of any type (e.g., collagen plugs, silicone plugs);
* History of intolerance or hypersensitivity to any component of the study medications;
* History or evidence of epithelial herpes simplex keratitis (dendritic keratitis); vaccinia; active or recent varicella viral disease of the cornea and/or conjunctiva; chronic bacterial disease of the cornea and/or conjunctiva and/or eyelids; mycobacterial infection of the eye; and/or fungal disease of the eye;
* Pregnant or lactating at the time of enrollment;
* Not willing to take adequate precautions not to become pregnant during the study;
* Use of any concomitant topical ocular medications during the study period;
* Use of systemic medications that may contribute to dry eye unless on a stable dosing regimen for a minimum of 30 days prior to Visit 1;
* Ocular conditions that may preclude the safe administration of either drop under investigation;
* Unwilling to discontinue contact lens wear during the study period and for at least 1 week prior to Visit 1;
* Participation in an investigational drug or device study within 30 days of entering this study;
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danyel C. Carr, MS, CCRA, Study Director — Alcon Research; Donald R Korb, O.D., Principal Investigator — Korb and Associates

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 1 study center located in the US.
Pre-assignment Details: This reporting group includes all subjects who were enrolled and received at least one of the study treatments (26).
Groups:
- Standard of Care: Microfiber towels (as warm compresses) warmed to the maximum comfortable temperature and placed over closed eyes for 8 minutes, 1 time a day. Duration of treatment was 3 months.
Period: Overall Study
Arm/Group | SYSTANE® Family | Standard of Care
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This reporting group includes all subjects who were enrolled and received at least one of the study treatments.
Groups:
- Total: Total of all reporting groups
Arm/Group | SYSTANE® Family | Standard of Care | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.1 (19.9) | 45.4 (19.8) | 41.7 (19.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Meibomian Glands Yielding Liquid Secretion (MGLYS)
Description: Meibomian gland functionality was evaluated by the investigator using the Meibomian Gland Evaluator (MGE), a handheld instrument that provides a standardized method for applying consistent, gentle pressure to the outer skin of the lower eyelid. The total number of meibomian gland orificies evidencing liquid secretion during expression with the MGE, in both eyes, was recorded. A lower number of functioning meibomian glands may contribute to dry eye syndrome.
Time Frame: Baseline, Month 1, Month 2, Month 3
Population: This reporting group includes all subjects who were enrolled and received at least one of the study treatments.
Measure: Mean (Standard Deviation); unit: functioning glands
Units Other Than Participants: Eyes
Arm/Group | SYSTANE® Family | Standard of Care
Number analyzed (Participants) | 13 | 13
Number analyzed (Eyes) | 26 | 26
functioning glands
  Baseline | 3.5 (1.50) | 4.2 (1.39)
  Month 1 | 7.0 (3.12) | 3.9 (1.76)
  Month 2 | 6.4 (2.45) | 3.5 (1.90)
  Month 3 | 9.3 (2.72) | 4.7 (2.29)

2. Secondary Outcome: Standard Patient Evaluation of Eye Dryness (SPEED) Questionnaire Responses
Description: The Standard Patient Evaluation of Eye Dryness (SPEED) Questionnaire is a 16-question validated questionnaire (resultant overall score 0-28, with 0 being best and 28 being worst) that measures the frequency and severity of dry eye symptoms. The SPEED questionnaire was completed by the patient with no assistance from the office staff, physician, or anyone else. Both eyes contributed to the mean.
Time Frame: Baseline, Month 1, Month 2, Month 3
Population: This reporting group includes all subjects who were enrolled and received at least one of the study treatments.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | SYSTANE® Family | Standard of Care
Number analyzed (Participants) | 13 | 13
Number analyzed (Eyes) | 26 | 26
units on a scale
  Baseline | 11.2 (2.59) | 11.2 (1.99)
  Month 1 | 8.2 (3.24) | 9.5 (3.91)
  Month 2 | 6.5 (3.02) | 7.9 (4.25)
  Month 3 | 5.0 (3.42) | 7.9 (4.46)

3. Secondary Outcome: Dry Eye Ocular Surface Disease Index (OSDI) Questionnaire Responses
Description: The Dry Eye OSDI Questionnaire is a 12-question validated questionnaire [resultant overall 0-100 score, with 0 being none of the time (best) and 100 being all of the time (worst)] that measures ocular symptoms, visual function, and environmental factors that may affect a patient's vision. The OSDI questionnaire was completed by the patient with no assistance from the office staff, physician, or anyone else. Both eyes contributed to the mean.
Time Frame: Baseline, Month 1, Month 2, Month 3
Population: This reporting group includes all subjects who were enrolled and received at least one of the study treatments.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | SYSTANE® Family | Standard of Care
Number analyzed (Participants) | 13 | 13
Number analyzed (Eyes) | 26 | 26
units on a scale
  Baseline | 32.3 (12.82) | 26.9 (15.42)
  Month 1 | 22.6 (10.48) | 21.0 (16.26)
  Month 2 | 16.1 (9.57) | 19.7 (17.42)
  Month 3 | 14.4 (10.20) | 17.9 (18.55)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of the study (4 months). This analysis group includes all enrolled and exposed subjects.
Description: An AE is defined as any untoward medical occurrence in a subject who is administered a study treatment (i.e., initiation of treatment with test article) regardless of whether or not the event has a causal relationship with the treatment. AEs were obtained through volunteered and elicited comments by the participant.
Arm/Group | SYSTANE® Family | Standard of Care
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 1/13 | 0/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SYSTANE® Family (N=13) | Standard of Care (N=13)
Infectious mononucleosis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.